CLINICAL TRIAL: NCT04687566
Title: Treatment Efficacy in Dextromethorphan, Memantine Monotherapy, or Combined Use of Dextromethorphan and Memantine in Patients With Amphetamine-type Stimulants Use Disorder
Brief Title: Dextromethorphan, Memantine Monotherapy, or Combined Use of Dextromethorphan and Memantine in Amphetamine Addiction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOST 109-2314-B-006-056
Record Dates: First submitted 2020-12-14; First posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Amphetamine Addiction; Pharmacotherapy
Keywords: amphetamine-type stimulants use disorder, dextromethorphan, memantine, inflammation, neurodegeneration, functional magnetic resonance imaging
MeSH Terms: conditions — Amphetamine-Related Disorders; Inflammation; Nerve Degeneration | interventions — Dextromethorphan; Memantine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- dextromethorphan (Experimental): Dextromethorphan, 60 mg per day, once daily, for 12 weeks
  Interventions: Drug: Dextromethorphan
- memantine (Experimental): Memantine, 5 mg per day, once daily, for 12 weeks
  Interventions: Drug: Memantine
- dextromethorphan and memantine (Experimental): Dextromethorphan (60mg per day) and memantine (5 mg per day) combination, once daily, for 12 weeks
  Interventions: Drug: Dextromethorphan and memantine
- placebo (Placebo Comparator): placebo, once daily, for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan — The participants will take dextromethorphan 60 mg per day, once daily, for 12 weeks. The participants will be blind to the assigned treatment group.
  Arms: dextromethorphan
Drug: Memantine — The participants will take memantine 5 mg per day, once daily, for 12 weeks. The participants will be blind to the assigned treatment group.
  Arms: memantine
Drug: Dextromethorphan and memantine — The participants will take dextromethorphan (60 mg per day) and memantine (5 mg per day) combination, once daily, for 12 weeks. The participants will be blind to the assigned treatment group.
  Arms: dextromethorphan and memantine
Drug: Placebo — The participants will take the placebo pills, once daily, for 12 weeks. The participants will be blind to the assigned treatment group.
  Arms: placebo

SUMMARY:
The investigators will conducted a randomized double-blind placebo-controlled study to investigate the treatment outcomes of add-on low dose dextromethorphan (DM), memantine (MM), or dextromethorphan and memantine combination (DM+MM) in amphetamine-type stimulants use disorder patients.

DETAILED DESCRIPTION:
The investigators will conducted a randomized double-blind placebo-controlled study to investigate the treatment outcomes of add-on low dose dextromethorphan (60mg/day, DM), memantine (5 mg/day, MM), or dextromethorphan (60mg/day) and memantine (5mg/day) combination (DM+MM) in amphetamine-type stimulants use disorder patients. The investigators will recruit 120 patients with ATSUD in three years and allocate participants to add-on DM, MM, DM+MM or placebo group in a 1:1:1:1 ratio (participants will also undergo usual psychosocial interventions).The investigators will follow up the participants for 12 weeks and measure the treatment responses, urine drug tests, craving scales and side effects to evaluate the therapeutic effects of add-on DM, MM, or DM+MM. Neuropsychological assessments, tests for inflammatory parameters and neurotrophic factors, and brain functional magnetic resonance imaging (fMRI) will also be evaluated during 12-weeks follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent by patient or legal representative.
2. Male or female patient aged ≧20 and ≦65 years.
3. A diagnosis of ATSUD according to DSM criteria made by a specialist in psychiatry.
4. Patient or a reliable caregiver can be expected to ensure acceptable compliance and visit attendance for the duration of the study.

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

1. Women of childbearing potential, not using adequate contraception as per investigator judgment or not willing to comply with contraception for the duration of the study.
2. Females who are pregnant or lactation.
3. Other major Axis-I DSM-IV diagnosis other than ATSUD, except for tobacco use disorder, ATS induced mood or psychotic disorders.
4. Current evidence of an uncontrolled and/or clinically significant medical condition, e.g., cardiac, hepatic and renal failure that would compromise patient safety or preclude study participation.
5. History of allergy or intolerable side effects of DM or MM.
6. Suicidal attempts or risks during screen or study period.
7. Presence of active infectious or autoimmune disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Urinary amphetamine positive rates | 12 weeks
  The urinary amphetamine tests will be examined during the 12 weeks of treatment period in patients with ATSUD and the results will be compared between the experimental and placebo groups.

SECONDARY OUTCOMES:
The Wisconsin Card Sorting Test (WCST) | 12 weeks
  The Wisconsin Card Sorting Test (WCST) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. Performance on the WCST was scored in terms of the total number of errors (TNE, range form 0-128), perseverative errors (PE, range from 0-118), conceptual level responses (CLRs, range from 0-100%), number of categories completed (NCC, range form 0-12), and trials to complete the first category (TCC, range from 0-128). Higher scores indicate worse performance in TNE, PE, and TCC. Higher scores indicate better performance in CLRs and NCC.
The Continuous performance tests (CPT) | 12 weeks
  Recognition Delayed (ARDM, range from 55-145), General Memory (GM, range from 40-168), and Working Memory (WM, range from 45-156 ). Higher scores indicate better performance.
  The Continuous performance tests (CPT) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. The CPT produces a standard set of performance measures that include the number of errors of omission and errors of commission. (1) Errors of omission occur when the participant fails to respond to the target stimulus. The omission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance. (2) Errors of commission occur when the participant responds to a non-target (X) stimulus. The commission errors t-scores are ranged from 20-80 (0-100%). Higher scores indicated worse performance.
The Wechsler Memory Scale - third edition (WMS-III) | 12 weeks
  The Wechsler Memory Scale - third edition (WMS-III) will be measured in patients with ATSUD at the initial screen period and at the endpoint (after 12 weeks of treatment). We will compare the changes from screen period to the endpoint between experimental and placebo group. WMS-III composite scores were calculated for the eight standardized primary indices: Auditory Immediate (AIM, range from 50-156), Visual Immediate (VIM, range from 47-162 ), Immediate Memory (IM, range from 40-164 ), Auditory Delayed (ADM, range from 46-162), Visual Delayed (VDM, range from 43-156), Auditory Recognition Delayed (ARDM, range from 55-145), General Memory (GM, range from 40-168), and Working Memory (WM, range from 45-156 ). Higher scores indicate better performance.
inflammatory markers | 12 weeks
  The plasma levels of cytokines and neurotrophic factors, tumor necrosis factor α (TNF-α[pg/mL]), C-reactive protein(CRP[pg/mL]), transforming growth factor β1 (TGF-β1 [pg/mL]), interleukin 6( IL-6[pg/mL]), interleukin 8(IL-8[pg/mL]), interleukin 1β (IL-1β[pg/mL]), and brain-derived neurotrophic factor(BDNF[pg/mL]), will be measured in patients with ATSUD at the initial screen period, day 1(baseline), week 4, 8, and 12(endpoint). We will compare the changes from screen period to the endpoint between the experimental and placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Yun Wang, Principal Investigator — National Cheng-Kung University Hospital
Locations (1):
- Department of Psychiatry, National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided